CLINICAL TRIAL: NCT00031109
Title: An Open-Label, Passive Antibody Trial to Assess Efficacy in the Pathogenic SHIV-89.6P Macaque Model of Human Antibodies Generated by a Candidate HIV-1 Vaccine in a Phase I Clinical Trial
Brief Title: The Effectiveness of Human Antibodies in Influencing an AIDS-Like Disease in Monkeys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: HVTN 803; 11636 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2002-02-25; First posted 2002-02-26 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Antibodies; HIV-1; HIV Envelope Protein gp160; Adjuvants, Immunologic; AIDS Vaccines; CD4 Lymphocyte Count; Disease Models, Animal; Antibody Formation; Macaca; Neutralization Tests; Viral Load; aluminum hydroxide; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Disease Models, Animal | interventions — Aluminum Hydroxide

INTERVENTIONS:
Biological: gp160 MN/LAI-2
Biological: Aluminum hydroxide

SUMMARY:
The purpose of this study is to see if an investigational vaccine can make antibodies (proteins found in blood) in humans that will influence the course of an AIDS-like disease in monkeys. Hopefully, the results of this study can be applied to humans.

AIDS, which is caused by infection with HIV, is associated with many deaths and occurrences of disease. Although recent advances have been made in anti-HIV therapy for AIDS, there is no cure for HIV infection or AIDS, and drug therapy is too expensive for most infected populations. Some organizations are trying to make safe and effective vaccines that may prevent HIV infection and AIDS worldwide. Certain vaccines can generate specific antibodies in humans, but they do not inhibit HIV infection in laboratory tests. It is possible, however, that these antibodies may make HIV disease less severe following infection. For this reason, monkeys will be used to evaluate the role of specific human antibodies.

DETAILED DESCRIPTION:
AIDS, caused by infection with the human immunodeficiency virus type 1 (HIV-1) is associated with enormous morbidity and mortality worldwide. Although recent advances have been made in antiretroviral therapy for AIDS, there is no cure for HIV infection or AIDS, and drug therapy is too expensive for most infected populations. The development of safe, effective vaccines to prevent HIV infection and AIDS worldwide is a commitment of some health-oriented organizations. A major goal in the effort to design an effective vaccine has been the identification of the immunologic correlates of protective immunity. Non-neutralizing antibodies might possess clinically important anti-HIV activities that remain to be defined and warrant investigation. The role played by antibody with minimal neutralizing activity induced by various HIV vaccination strategies is unknown. It is possible that low-level neutralization or other activities may lead to an improvement or worsening in disease course following infection. For this reason it is proposed that a challenge trial in the rhesus macaque SHIV model be performed, in which the role of such antibodies, which are derived from non-infected human vaccinees, will be evaluated.

This is a 2-part study. Part I involves human participants; Part II involves rhesus macaques.

Part 1: Human participants are divided into 2 groups:

Group I: Participants who previously were enrolled in specific AIDS Vaccine Evaluation Group (AVEG) protocols are immunized with a single dose of the recombinant gp160MN/LAI-2 vaccine in alum (aluminum hydroxide adjuvant) on Day 0 of the study.

Group II: Participants who are vaccine naive receive no immunization. Each participant will have 5 clinic visits during the study. Blood is drawn at each visit for routine testing and immune system check. Sera is drawn from participants for neutralizing antibody determination. Approximately 3 weeks after immunization (Day 18), blood is drawn from participants of both groups for a plasmapheresis procedure in which platelets and plasma are removed. This process is repeated 1 week later. Immunoglobulin G (IgG) is purified from the plasma of vaccinated participants.

Part II: Juvenile rhesus macaques are divided into 4 groups and are infused with IgG from human participants of Groups I and II at Day 0. At Day 1, the macaques are exposed to SHIV-89.6P. At Days 3, 7, 10, and weekly up to Day 73, the CD4 lymphocyte count, plasma viremia, and antibodies of the macaques are measured.

ELIGIBILITY:
Inclusion Criteria

Participants in Groups I and II may be eligible for this study if they:

* Are in good general health.
* Have a negative HIV blood test within 8 weeks prior to enrollment.
* Agree to use acceptable methods of contraception for at least 21 days prior to enrollment until the last protocol visit, if a woman is participating in sexual activity that could lead to pregnancy. A woman who cannot have children, is not sexually active, or whose male partner(s) has undergone successful vasectomy does not have to use contraception.
* Have access to a participating HIV vaccine trials unit (HVTU) and are willing to be followed for 4 months, the planned study duration.
* Participants in Group I may be eligible for this study if they:
* Have participated in AVEG trial 022, 022A, 026, 029, or 202 and received full immunization schedule of ALVAC-HIV (vCP205 or vCP300) and HIV-1 SF-2 rgp120 combination.
* Have a peak concentration of neutralizing antibody to MN greater than 1:800 during AVEG 022, 022A, 026, 029, or 202.
* Participants in Group II may be eligible for this study if they:
* Are 18-60 years old.

Exclusion Criteria

Participants in Groups I and II may not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have received live attenuated vaccines within 30 days prior to enrollment.
* Have received certain vaccines (e.g., flu, pneumococcal, allergy) within 14 days of study vaccine administration.
* Have used investigational research agents within 30 days prior to enrollment.
* Have received HIV vaccines or placebo in a vaccine trial. Note: not required for participants in Group I.
* Have received blood products within 120 days prior to HIV screening.
* Have received immunoglobulin within 60 days prior to HIV screening.
* Have had serious harmful reactions to vaccines.
* Have immunodeficiency or autoimmune disease.
* Have cancer.
* Have taken (within the last 6 months) or are currently taking immunosuppressive drugs.
* Have type I or type II diabetes mellitus including cases controlled with diet alone.
* Have a thyroid disease including thyroidectomy and diagnoses requiring drugs.
* Have unstable asthma.
* Are taking anti-tuberculosis (TB) prophylaxis or therapy.
* Have a seizure disorder.
* Have a bleeding disorder diagnosed by a doctor.
* Have had a splenectomy.
* Have serious angioedema.
* Have active syphilis.
* Have high blood pressure.
* Have a mental condition that will affect their participation in the protocol.
* Have any clinically significant condition for which plasmapheresis would pose additional risk to the participant.
* Participants in Group I may not be eligible for this study if they:
* Have received an HIV vaccine or placebo in a vaccine trial other than AVEG 022, 022A, 026, 029, or 202.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Evans, Study Chair; Sharon Frey, Study Chair

REFERENCES:
- [Background] Evans TG, Frey S, Israel H, Chiu J, El-Habib R, Gilbert P, Gaitan A, Montefiori DC; HIV Vaccine Trials Network (HVTN 803). Long-term memory B-cell responses in recipients of candidate human immunodeficiency virus type 1 vaccines. Vaccine. 2004 Jun 30;22(20):2626-30. doi: 10.1016/j.vaccine.2003.12.011. PMID 15193388